CLINICAL TRIAL: NCT07006428
Title: Visual Performance Differences Between Clareon PanOptix and a Comparable Multifocal Intraocular Lens
Brief Title: Visual Performance of Clareon PanOptix vs. a Comparable Multifocal Intraocular Lens
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Argus Research Center, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUPER-IIT-96028407
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Age Related Cataracts
Keywords: Clareon PanOptix; Multifocal IOL; Cataract Surgery; Visual Acuity; Intraocular Lens

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Clareon PanOptix or PanOptix Toric IOLs (Experimental)
  Interventions: Device: Clareon PanOptix or PanOptix Toric IOLs
- Comparable multifocal IOL (Experimental)
  Interventions: Device: Comparable multifocal IOL

INTERVENTIONS:
Device: Clareon PanOptix or PanOptix Toric IOLs — Bilateral implantation of the Clareon PanOptix or PanOptix Toric IOLs.
  Arms: Clareon PanOptix or PanOptix Toric IOLs
Device: Comparable multifocal IOL — Bilateral implantation of a comparable multifocal IOL
  Arms: Comparable multifocal IOL

SUMMARY:
This is a two-part, multi-center, investigator-initiated clinical study comparing visual outcomes and patient satisfaction in subjects receiving bilateral implantation of either the Clareon PanOptix intraocular lens (IOL) or a comparable multifocal IOL. The study includes a retrospective/prospective pilot phase and a prospective, randomized comparison phase.

ELIGIBILITY:
Inclusion Criteria:

Stage 1: IIT Pilot

* Willing and able to understand and sign informed consent.
* Adult patients previously diagnosed with age-related cataracts bilaterally.
* Previous bilateral age-related cataract removal and with bilateral implantation of the Clareon PanOptix/ Clareon PanOptix Toric (T3-T4) or Comparable Multifocal Intraocular Lens (equivalent to T3-T4) closest to 2.5-5-months after implantation and >2 weeks post YAG (if done) that were targeted for emmetropia.
* Best monocular corrected distance visual acuity was expected to be 0.1 logMAR (Snellen 20/25) or better in both eyes pre-operatively as determined by surgeon.
* Normal ocular findings aside from cataract.

Stage 2: Comparison

* Willing and able to understand and sign informed consent.
* Adult patient diagnosed with age-related cataracts bilaterally.
* Planned bilateral cataract removal by femtosecond laser-assisted phacoemulsification with bilateral implantation of the Clareon PanOptix/Clareon PanOptix Toric (T3-T4) or Comparable Multifocal Intraocular Lens (equivalent to T3-T4).
* Best monocular corrected distance visual acuity expected to be 0.1 logMAR (Snellen 20/25) or better in both eyes postoperatively as determined by surgeon.
* Residual astigmatism expected to be ≤ 0.50 diopters in both eyes postoperatively as determined by surgeon (after using either toric IOL or arcuate incision with laser).
* Normal ocular findings aside from cataract.

Exclusion Criteria:

Stage 1: IIT Pilot

* Corneal pathology, irregular astigmatism, preexisting macular disease and other retinal degenerative diseases, diabetic retinopathy that is expected to cause future vision loss, glaucoma, severe dry eye disease, nystagmus, strabismus, zonular laxity or dehiscence, pseudoexfoliation.
* Previous history of any ocular surgery including corneal refractive surgery.
* Participation in another clinical study that could interfere with the results.
* Patients with monovision correction.
* Any active ocular infection or inflammation.

Stage 2: Comparison

* Corneal pathology, irregular astigmatism, preexisting macular disease and other retinal degenerative
* diseases that is expected to cause future vision loss, glaucoma, severe dry eye disease, nystagmus, strabismus, zonular laxity or dehiscence, pseudoexfoliation.
* Previous history of any ocular surgery including corneal refractive surgery.
* Participants desiring monovision.
* History of amblyopia or monofixation syndrome with poor stereoscopic vision.
* Total corneal HOA greater than 0.6um, coma less than 0.3um at 4mm-5mm scan depending on pre- op photopic topography.
* Any planned simultaneous/combined procedures at time of cataract surgery (e.g. MIGs).
* Participation in another clinical study that could interfere with the results.
* Any active ocular infection or inflammation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Binocular photopic BCDVA (4m) | 2.5 to 5 months postoperatively
Binocular BCDVA (4m) | Month 3

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Tyson Eye, Cape Coral, Florida
  - North Georgia Eye Associates, Gainesville, Georgia

IPD SHARING:
Plan to Share IPD: No